CLINICAL TRIAL: NCT06300216
Title: A Real-world Study of Octreotide Microspheres in Chinese Patients With Neuroendocrine Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202401-034-1
Record Dates: First submitted 2024-02-25; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-02

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Octreotide microspheres standard dose monotherapy
  Interventions: Drug: Octreotide microspheres
- Octreotide microspheres standard dose combination therapy
- Octreotide microspheres incremental or increased frequency therapy
- Octreotide microspheres maintenance therapy after targeted or chemotherapy

INTERVENTIONS:
Drug: Octreotide microspheres — 20mg/30mg Q4W
  Groups: Octreotide microspheres standard dose monotherapy

SUMMARY:
The aim of this multicenter, open-label, observational study is to evaluate the safety and efficacy of octreotide microspheres in the treatment of advanced neuroendocrine tumors in real clinical practice, especially to evaluate the treatment of octreotide microspheres in various subgroups of neuroendocrine tumor patients.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an informed consent form and voluntarily participate in this study;
2. Patients with unresectable or metastatic neuroendocrine tumors confirmed by histopathology. Patients with recurrence and progression after surgery or local treatment can also be included in the study;
3. Age ≥ 18 years old;
4. Treatment with octreotide microspheres.

Exclusion Criteria:

1. Confirmed pregnant or lactating women;
2. Participating in any research with intervention measures outside of routine clinical practice;
3. Other situations unsuitable for inclusion in the study determined by the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced neuroendocrine tumors treated with octreotide microspheres will be eligible to participate in the study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03-26 (Estimated); Primary Completion 2027-11-26 (Estimated); Study Completion 2028-05-26 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events | up to 46 months
  Treatment emergent adverse events were recorded according to Common Terminology Criteria for Adverse Events (version 5.0) of the National Cancer Institute that participants received at least one dose of protocol treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Hao, Dr., Principal Investigator — Qilu hospital of Shandong University, China
Locations (1):
- Qilu hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No